CLINICAL TRIAL: NCT05039138
Title: EFFECT OF NEUROMUSCULAR TRAINING ON SHOULDER FUNCTION IN PATIENTS WITH SHOULDER IMPINGEMENT SYNDROME: A DOUBLE BLINDED RANDOMIZED CONTROLLED TRIAL
Brief Title: EFFECT OF NEUROMUSCULAR TRAINING ON SHOULDER FUNCTION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Ahmed Elnour Noaman Nada, researcher, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: shoulder neuromuscular
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: NMT
Keywords: NMT= NEUROMUSCULAR TRAINING

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (control) (Experimental): : it includes 17 patients who will receive traditional strength training program.
  Interventions: Other: traditional training exerises
- Group II (experimental): (Experimental): it includes 17 patients who will receive upper extremity neuromuscular training exercises
  Interventions: Other: NEUROMUSCULAR TRAINING EXERCISE

INTERVENTIONS:
Other: NEUROMUSCULAR TRAINING EXERCISE — patients will receive neuromuscular training exercises in group II
  Arms: Group II (experimental):
Other: traditional training exerises — traditional strength training exercises in group I
  Arms: Group I (control)

SUMMARY:
This study will be conducted to compare the effect of neuromuscular training versus traditional strength training in terms of shoulder joint function, proprioception accuracy and isometric external and internal rotator muscles strength in patients with SIS, it will be conducted at the out-patient clinic of physical therapy in Pharos University in Alexandria, Egypt

DETAILED DESCRIPTION:
Double-blinded randomized controlled trial (patient and research assistant (the examiner of all patients) will be blinded).

Participants:

Thirty-four patients of both genders will be selected through non-probability sampling diagnosed as Neer's stage II SIS and their age range from 25-45 years will be randomly assigned to 1 of 2 groups. Each patient will sign an informed consent before starting the study (Appendix III).

Eligible patients will be recruited by physical therapist via referral from the treating orthopedic surgeon who will diagnose SIS based on clinical and radiological examination.

Group I (control): it includes 17 patients who will receive traditional strength training program.

Group II (experimental): it includes 17 patients who will receive upper extremity neuromuscular training exercises

ELIGIBILITY:
Inclusion Criteria:

* Patient age from 25-40 with a clinical diagnosis of Neer's stage II SIS (Consigliere et al., 2018).

Shoulder pain for at least three months (Heron et al., 2017) Painful arc of movement during flexion or abduction (Heron et al., 2017). Positive Neer's or Kennedy- Hawkins Test (Heron et al., 2017). Pain on resisted external rotation, abduction or Empty Can Test (Ager et al., 2019).

Exclusion Criteria:

Symptoms of cervical radiculopathy. Diagnosed inflammatory disorder. Neurological disorder. Widespread pain condition. Evidence of complete RC tear (positive drop arm test). Previous surgery to the affected shoulder.

:

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-12-20 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
SPADI (The Shoulder Pain and Disability Index) | 6 weeks
  It is a self-report questionnaire for shoulder function
Inclinometer | 6 weeks
  joint position sense
Hand held dynamometer | 6 weeks
  isometric muscle strength

IPD SHARING:
Plan to Share IPD: Undecided